CLINICAL TRIAL: NCT04685460
Title: Clinical Study of 3D Printed Bolus for Volumetric Modulated Arc Therapy of Post-mastectomy Treatment
Brief Title: 3D Printed Bolus in Post-mastectomy Radiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: jcl2020-2 breast cancer
Record Dates: First submitted 2020-11-18; First posted 2020-12-28 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2020-11

CONDITIONS: Breast Neoplasms; Radiotherapy Side Effect
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D-printed bolus (Experimental)
  Interventions: Other: customized 3D-printed bolus fabricated based on reconstruction of computed tomography (CT) images
- Conventional bolus (No Intervention)

INTERVENTIONS:
Other: customized 3D-printed bolus fabricated based on reconstruction of computed tomography (CT) images — customized 3D-printed bolus fabricated based on reconstruction of computed tomography (CT) images were used in this study.
  Arms: 3D-printed bolus

SUMMARY:
Recently, there is growing interest in the application of three-dimensional (3D) printed bolus to radiotherapy.At present, the researches on the application of 3D-printed bolus in breast cancer are mainly focused on air gap between skin and bolus or electron beam conformal therapy [7,15], there are no clinical experience with customized 3D-printed bolus for volumetric modulated arc therapy (VMAT) in daily practice has been published up to now. We aim to evaluate dosimetry and application of 3D-printed bolus for the post-mastectomy radiotherapy (PMRT) with Volumetric modulated arc therapy (VMAT). Seventy five patients with breast cancer receiving radiotherapy following post-mastectomy in our department were randomly selected in this study. The accuracy of fit of the 3D-Printed bolus to the chest wall was improved significantly relative to conventional bolus.This study demonstrates customized 3D-printed bolus in post-mastectomy radiation therapy improves fit of the bolus compared to conventional bolus. Furthermore, VMAT based on 3D-printed bolus significantly improves the chest wall target coverage and the conformity of plan, and reduces the dose of ipsilateral lung and heart, compared to conventional bolus.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer patients with post-mastectomy treatment

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-20 (Estimated)

PRIMARY OUTCOMES:
dose comparison | one year
  The prescription dose was 50 Gy in 25 fractions. Dose-volume histograms (DVHs) were used dosimetric analysis. D98%, D50% and D2%, indicating dose to 98% (near-minimum dose), 50% and 2% (near-maximum dose) of both target volumes, and V95%, V100%, and V110% indicating percent volume receiving 95%, 100% and 110% of prescribed dose, were recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangxi Cancer Hospital of Nanchang University, Nanchang, Jiangxi, China